CLINICAL TRIAL: NCT01968473
Title: An Evaluation of Comfort and Tolerance of Surface Neuro Muscular Electrical Stimulation (NMES), When Applied to Parkinson's Disease Patients for Both Sensory and Motor Activation.
Brief Title: Comfort and Tolerance of Surface Neuro Muscular Electrical Stimulation in Parkinson's Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Gearoid O Laighin, Professor, National University of Ireland, Galway, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: NMES_PD_Comfort
Record Dates: First submitted 2013-09-09; First posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Freezing of Gait; Neuromuscular Electrical Stimulation; Comfort; Pain tolerance; Pain; Sensory threshold; Motor threshold; Pain threshold
MeSH Terms: conditions — Parkinson Disease; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NMES Device comfort (Experimental): NMES Device comfort, establishing Sensory, Motor and Pain thresholds. Max Pain tolerance is also established.
  Interventions: Device: NMES Device comfort

INTERVENTIONS:
Device: NMES Device comfort — NMES device, establishing Sensory, Motor and Pain thresholds and Pain tolerance.
  Other Names: Device name: Duo-Stim

SUMMARY:
The purpose of this study is to investigate issues relating to comfort and tolerance to surface neuro muscular electrical stimulation in a parkinson disease population.

DETAILED DESCRIPTION:
The comfort and tolerance of Parkinson Disease (PD) patients to surface neuro muscular electrical stimulation (NMES) will be investigated.

Six muscle sites will be tested sensory, motor and pain thresholds recorded. Furthermore pain tolerance will be recorded as the level at which the stimulus is unbearable.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic PD (UK, PD Brain Bank Criteria)
* A Hoehn and Yahr stage of 2 - 4
* Exhibiting Freezing of Gait or another gait abnormalityin the ON or OFF state.
* An ability to mobilise independently for the purpose of research when in the 'off' state
* An ability to walk unaided for 10 meters.

Exclusion Criteria:

* A serious cognitive impairment (MMSE<24)
* Pregnant or currently involved in another clinical trial.
* Uncontrolled heart problems
* Pacemakers
* On opioid or neuropathic pain medication

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Patient comfort in response to neuromuscular electrical stimulation in Parkinson's disease. | 1 day
  Participants will be tested over a range of stimulation intensities at different muscle sites. Primary outcome measure will be patient comfort and tolerance to neuromuscular electrical stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Gearoid O'Laighin, PhD, Principal Investigator — Electrical & Electronic Engineering NUI Galway
Locations (1):
- University Hospital Galway, Galway, Ireland